CLINICAL TRIAL: NCT05262179
Title: A Phase 1 Clinical Trial to Explore Systemic Exposure of CTO0101 Eye Drops, Safety and Local Tolerability in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTO0101
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTO0101 (Experimental)
  Interventions: Drug: CTO0101
- Placebo (Vehicle) (Placebo Comparator)
  Interventions: Other: Placebo (vehicle)

INTERVENTIONS:
Drug: CTO0101 — 1 drop/ once or three times a day/ for 17 days divided into stage2
  Arms: CTO0101
Other: Placebo (vehicle) — 1 drop/ once or three times a day/ for 17 days divided into stage2
  Arms: Placebo (Vehicle)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetic characteristic of CTO0101

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers
* Written informed consent to participate in the trial

Exclusion Criteria:

* Those who have a history of ophthalmic diseases and surgery within 5 years
* Smokers with an average daily smoking amount exceeding 10 cigarettes

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-05-27 (Estimated); Study Completion 2022-07-05 (Estimated)

PRIMARY OUTCOMES:
Cmax,ss | Day8 of stage 2
Tmax,ss | Day8 of stage 2
t1/2,ss | Day8 of stage 2
AUCτ,ss | Day8 of stage 2
RAAUCτ | Day8 of stage 2

CONTACTS AND LOCATIONS:
Locations (1):
- Taejoon Pharmaceutical Co., Ltd., Seoul, South Korea